CLINICAL TRIAL: NCT05830396
Title: GRoningen Early-PD Ambroxol Treatment (GREAT) Trial: A Randomised, Double-blind, Placebo-controlled, Singlecenter Trial With Ambroxol in Parkinson Patients With a GBA Mutation
Brief Title: GRoningen Early-PD Ambroxol Treatment
Acronym: GREAT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202100266
Record Dates: First submitted 2023-03-20; First posted 2023-04-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Parkinson; Parkinson Disease
Keywords: Ambroxol; GBA1; GBA
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambroxol (Experimental): Ambroxol 1800mg/day
  Interventions: Drug: Ambroxol Hydrochloride
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambroxol Hydrochloride — Patients will either receive ambroxol or placebo. ambroxol will be given intially in a dosage of 600mg/day. After 1 week, this will be increased to 1200mg/day. After 2 weeks the maximum dosage of 1800mg/day will be given. In total, ambroxol will be administered for 48 weeks. This is followed by a 12 week washout period, after wich the final outcomes will be measured (week 60).
  Arms: Ambroxol
Drug: Placebo — Patients will either receive ambroxol or placebo. ambroxol will be given intially in a dosage of 600mg/day. After 1 week, this will be increased to 1200mg/day. After 2 weeks the maximum dosage of 1800mg/day will be given. In total, ambroxol will be administered for 48 weeks. This is followed by a 12 week washout period, after wich the final outcomes will be measured (week 60).
  Arms: Placebo

SUMMARY:
The most common genetic risk factor for Parkinson's Disease is a heterozygous mutation of the GBA1 gene, encoding the lysosomal enzyme glucocerebrosidase (GCase). Reduced GCase activity is associated with aggregation of the protein alpha synucleine (aSyn) in the central nervous system, which is related to the pathological cause of PD. Ambroxol is a mucolytic expectorant that appears to facilitate the refolding of the misfolded GBA protein thats acts as a chaperone for GCase.

This randomized placebo-controlled trial aims to investigate the disease-modifying properties of ambroxol in PD patients with a GBA1-mutation. Patients will undergo motor and cognitive tests, as well as imaging and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease, according to Movement Disorders Society (MDS) criteria (27)
* Disease duration of 10 years or less at time of inclusion
* PD patients carrying a GBA1 mutation
* Able to write written informed consent, understanding study protocol and perform protocol related actions
* Willing and able to self-administer oral ambroxol or placebo medication

Exclusion Criteria:

* The refusal to be informed about an unforeseen clinical finding
* Use of an implanted Deep Brain Stimulation (DBS) system
* Confirmed dysphagia that would preclude self-administration of ambroxol or placebo tablets
* History of known sensitivity to the study medication
* Pregnant or breastfeeding women
* Participants of childbearing potential that would not use adequate birth control, consisting of a negative pregnancy test at the screening visit and use of accepted contraceptive methods defined as highly effective while participating in the study
* MRI incompatible implants in the body
* Any clinically significant or unstable medical or surgical condition that in the opinion of the principal investigator may put the participant at risk when participating in the study or may influence the results of the study or affect the participant's ability to take part in the study, as determined by medical history, physical examinations, electrocardiogram (ECG), or laboratory tests. Such conditions may include:

  1. Impaired renal function (a positive urine dipstick test, and laboratory values below or above: a eGFR <45 ml/min 1,73M2, Sodium 135-145 mmol/L, Potassium 3.5-5.0 mmol/L, Urea 2.5-7.5mmol/L).
  2. Moderate/severe hepatic impairment (laboratory values below or above: ASAT 0- 80U/L, ALAT0-90 U/L, GGT > 80 U/L, Alkaline Phosphatase 35-210 U/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS3 motor scale | 60 weeks
  Motor scale developed for PD patients, 0-132. 0 means good performance, 132 means very bad performance

SECONDARY OUTCOMES:
Safety and tolerability measured by incidence of adverse events and possible side effects | all throughout the study. specifically at: 1, 2, 3, 12, 24, 36, 48, 60 weeks
  AE will be monitored and patients will be questioned about side effects every week during the first 3 weeks and after that, every 3 months during the visits
Glucocerebrosidase (GCase) activity in blood mononuclear cells | 0, 12, 60 weeks
  Measured by the level of sphingolipids in PBMCs
Striatal F-DOPA uptake as measured by [18] F-DOPA PET scan | 0, 60 weeks
fMRI resting state to investigate the functional architecture and structural MRI for PET-scan | 0, 60 weeks
  Fluctuations in the BOLD signal can be used to investigate the functional architecture and connectivity within the brain.
Quality of Life (PDQ-39 questionnaire) | 0, 60 weeks
Non Motor Symptoms (NMSS scale) | 0, 60 weeks
  minimum value is 0, maximum value is 360. 0 indicating a good performance, 360 indicating a very bad performance
Cognition, using the Montreal Cognitive Assessment (MoCA) | 0, 60 weeks
  Range is 0-30, 0 indicating the worst performance, 30 indicating the best performance

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siemeling O, Slingerland S, van der Zee S, van Laar T. Study protocol of the GRoningen early-PD Ambroxol treatment (GREAT) trial: a randomized, double-blind, placebo-controlled, single center trial with ambroxol in Parkinson patients with a GBA mutation. BMC Neurol. 2024 May 1;24(1):146. doi: 10.1186/s12883-024-03629-9. PMID 38693511